CLINICAL TRIAL: NCT03349632
Title: Clinical Comparison of 4 Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C004
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Refractive Error
Keywords: Contact lenses; Myopia; Near-sighted; Daily disposable
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- DD T2/Oasys 1-Day (Other): Verofilcon A contact lenses and senofilcon A contact lenses worn in both eyes, each product, for 1 week on a daily wear basis, as randomized
  Interventions: Device: verofilcon A contact lenses; Device: senofilcon A contact lenses
- DD T2/MyDay (Other): Verofilcon A contact lenses and stenfilcon A contact lenses worn in both eyes, each product, for 1 week on a daily disposable basis, as randomized
  Interventions: Device: verofilcon A contact lenses; Device: stenfilcon A contact lenses
- DD T2/Moist (Other): Verofilcon A contact lenses and etafilcon A contact lenses worn in both eyes, each product, for 1 week on a daily disposable basis, as randomized
  Interventions: Device: verofilcon A contact lenses; Device: etafilcon A contact lenses

INTERVENTIONS:
Device: verofilcon A contact lenses — Investigational spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: DDT2
Device: senofilcon A contact lenses — Commercially available spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: ACUVUE OASYS® 1-Day with HydraLuxe™ Technology; Oasys 1-Day
  Arms: DD T2/Oasys 1-Day
Device: stenfilcon A contact lenses — Commercially available spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: MyDay®; MyDay
  Arms: DD T2/MyDay
Device: etafilcon A contact lenses — Commercially available spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: 1-Day ACUVUE® MOIST; Moist
  Arms: DD T2/Moist

SUMMARY:
The purpose of this study is to obtain on-eye performance data to inform contact lens product development and to further evaluate product performance in the intended population.

DETAILED DESCRIPTION:
The expected duration of subject participation in the study is approximately 20 days with 3 scheduled visits. Each subject will evaluate the test contact lenses compared to 1 of 3 commercially available contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and must sign an approved Informed Consent Form
* Successfully wears daily disposable spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months
* Best Corrected Visual Acuity of 20/25 Snellen or better in each eye
* Willing to stop wearing habitual contact lenses for the duration of study participation
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Any eye condition, surgery, disease, or use of medication that contraindicates contact lens wear, as determined by the Investigator.
* Routinely sleeps in habitual contact lenses
* Currently wears Oasys 1-Day, MyDay, or Moist contact lenses
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Pensacola, Florida
  - Alcon Investigative Site, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigational sites located in the United States.
Pre-assignment Details: Of the 68 enrolled, 2 subjects exited as screen failures prior to randomization. This reporting group includes all randomized subjects (66).
Groups:
- DD T2/Oasys 1-Day (Sequence 1): Verofilcon A contact lenses worn in Period 1, followed by senofilcon A contact lenses worn in Period 2. Each product worn bilaterally (in both eyes) for 1 week on a daily wear basis, as randomized
- Oasys 1-Day/DD T2 (Sequence 2): Senofilcon A contact lenses worn in Period 1, followed by verofilcon A contact lenses worn in Period 2. Each product worn bilaterally for 1 week on a daily wear basis, as randomized
- DD T2/MyDay (Sequence 3): Verofilcon A contact lenses worn in Period 1, followed by stenfilcon A contact lenses worn in Period 2. Each product worn bilaterally for 1 week on a daily wear basis, as randomized
- MyDay/DD T2 (Sequence 4): Stenfilcon A contact lenses worn in Period 1, followed by verofilcon A contact lenses worn in Period 2. Each product worn bilaterally for 1 week on a daily wear basis, as randomized
- DD T2/Moist (Sequence 5): Verofilcon A contact lenses worn in Period 1, followed by etafilcon A contact lenses worn in Period 2. Each product worn bilaterally for 1 week on a daily wear basis, as randomized
- Moist/DD T2 (Sequence 6): Etafilcon A contact lenses worn in Period 1, followed by verofilcon A contact lenses worn in Period 2. Each product worn bilaterally for 1 week on a daily wear basis, as randomized
Period: Period 1, First Week of Wear
Arm/Group | DD T2/Oasys 1-Day (Sequence 1) | Oasys 1-Day/DD T2 (Sequence 2) | DD T2/MyDay (Sequence 3) | MyDay/DD T2 (Sequence 4) | DD T2/Moist (Sequence 5) | Moist/DD T2 (Sequence 6)
Started | 11 | 11 | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2, Second Week of Wear
Arm/Group | DD T2/Oasys 1-Day (Sequence 1) | Oasys 1-Day/DD T2 (Sequence 2) | DD T2/MyDay (Sequence 3) | MyDay/DD T2 (Sequence 4) | DD T2/Moist (Sequence 5) | Moist/DD T2 (Sequence 6)
Started | 11 | 11 | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study (Safety Analysis Set).
Groups:
- Overall: Verofilcon A contact lenses with corresponding control product (senofilcon A, stenfilcon A, or etafilcon) worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56
  Black or African American | 6
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision
Description: Overall quality of vision was collected binocularly and rated on a 10-point scale with 1 = poor to 10 = excellent. Subjects were asked "Thinking back over the last week, please rate our study lenses. Rate eyes together." No formal hypotheses was conducted; hence no inferential testing was performed.
Time Frame: Day 8, each product
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DD T2 (Sequence 1 and 2); DD T2 (Sequence 3 and 4); DD T2 (Sequence 5 and 6): Verofilcon A contact lenses worn in Period 1 or Period 2 for 1 week
- Oasys 1-Day (Sequence 1 and 2): Senofilcon A contact lenses worn in Period 1 or Period 2 for 1 week
- MyDay (Sequence 3 and 4): Stenfilcon A contact lenses worn in Period 1 or Period 2 for 1 week
- Moist (Sequence 5 and 6): Etafilcon A contact lenses worn in Period 1 or Period 2 for 1 week
Arm/Group | DD T2 (Sequence 1 and 2) | Oasys 1-Day (Sequence 1 and 2) | DD T2 (Sequence 3 and 4) | MyDay (Sequence 3 and 4) | DD T2 (Sequence 5 and 6) | Moist (Sequence 5 and 6)
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22
units on a scale | 8.5 (1.4) | 9.2 (1.3) | 8.8 (1.8) | 9.4 (0.8) | 9.2 (1.1) | 8.8 (1.7)

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 2 weeks
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Safety Analysis Set, based on treatment-specific exposure.
Groups:
- Oasys 1- Day (Sequence 1 and 2): Senofilcon A contact lenses worn in Period 1 or Period 2 for 1 week
Arm/Group | DD T2 (Sequence 1 and 2) | Oasys 1- Day (Sequence 1 and 2) | DD T2 (Sequence 3 and 4) | MyDay (Sequence 3 and 4) | DD T2 (Sequence 5 and 6) | Moist (Sequence 5 and 6)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT03349632/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03349632/SAP_001.pdf